CLINICAL TRIAL: NCT07397208
Title: Assessment of the Repeatability of Sublingual Microcirculation Function Measurements in Healthy Volunteers and Critically Ill Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Other Study IDs: MICRO-powt
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Critical Illness; Healthy
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Healthy Volunteers
- Critically ill: Patients Hospitalized in the ICU

SUMMARY:
The assessment of microcirculatory function plays a pivotal role in perioperative medicine and intensive care. One promising method for evaluating microcirculatory function is the microscopic analysis of the oral mucosal microvasculature. However, this method is not currently fully validated.

The aim of this study is to assess the repeatability of sublingual microcirculation measurements using the CytoCam-IDF device (Braedius Medical).

ELIGIBILITY:
Group 1: Healthy Volunteers

Inclusion Criteria:

* ASA Physical Status I-II
* Age 18-40 years

Exclusion Criteria:

* Chronic diseases
* Chronic medication use
* Pregnancy
* Use of stimulants (caffeine, nicotine, alcohol) within 12 hours prior to the study
* Lack of consent to participate

Group 2: Patients Hospitalized in the ICU

Inclusion Criteria:

* Age > 18 years
* Hospitalization in the Intensive Care Unit (ICU)
* Requirement for vasoactive drugs (minimum norepinephrine equivalent dose >0.1μg/kg / min )
* Mechanical ventilation via an endotracheal tube

Exclusion Criteria:

* Head and craniofacial trauma
* Pregnancy
* Intensive fluid therapy (>200ml/h)
* Changes in vasoactive drug dosages within 30 minutes prior to study inclusion
* Hypothermia (body temperature <35.5 oC)
* Fever (body temperature >38.5oC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the ICU at the University Clinical Center in Gdańsk, or healthy volunteers
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02-07 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
FCD (Functional Capillary Density) | From enrollment every 5 minutes (3 measurements per operator) - approx. 20 min.
  Sublingual Microcirculation Assessment Sublingual microcirculation will be assessed using the CytoCam-IDF camera (Braedius Medical, Huizen, The Netherlands). The measurement technique involves gently applying the microscope probe with a disposable cap to the sublingual mucosa and recording short video sequences. The device utilizes green LED light to visualize moving blood cells, allowing for subsequent computerized analysis of capillary density and flow quality within the microvessels. Two operators will perform 3 series of measurements at 5-minute intervals with Cytocam - IDF microcirculation camera. Each series will consist of measurements taken from 3 adjacent sites. All measurements will be performed by the same two individuals
  Unit of measurement: mm/mm^2
MFI (Microvascular Flow Index) | From enrollment every 5 minutes (3 measurements per operator) - approx. 20 min.
  Sublingual Microcirculation Assessment Sublingual microcirculation will be assessed using the CytoCam-IDF camera (Braedius Medical, Huizen, The Netherlands). The measurement technique involves gently applying the microscope probe with a disposable cap to the sublingual mucosa and recording short video sequences. The device utilizes green LED light to visualize moving blood cells, allowing for subsequent computerized analysis of capillary density and flow quality within the microvessels. Two operators will perform 3 series of measurements at 5-minute intervals with Cytocam - IDF microcirculation camera. Each series will consist of measurements taken from 3 adjacent sites. All measurements will be performed by the same two individuals
  Unit of measurement: 0 - no flow / 1 -intermittent flow / 2 - sluggish flow / 3 - continuous flow
HI (Heterogeneity Index) | From enrollment every 5 minutes (3 measurements per operator) - approx. 20 min.
  Sublingual Microcirculation Assessment Sublingual microcirculation will be assessed using the CytoCam-IDF camera (Braedius Medical, Huizen, The Netherlands). The measurement technique involves gently applying the microscope probe with a disposable cap to the sublingual mucosa and recording short video sequences. The device utilizes green LED light to visualize moving blood cells, allowing for subsequent computerized analysis of capillary density and flow quality within the microvessels. Two operators will perform 3 series of measurements at 5-minute intervals with Cytocam - IDF microcirculation camera. Each series will consist of measurements taken from 3 adjacent sites. All measurements will be performed by the same two individuals
  Unit of measurements none, relative measurement

SECONDARY OUTCOMES:
TVD (Total Vessel Density) | From enrollment every 5 minutes (3 measurements per operator) - approx. 20 min.
  Sublingual Microcirculation Assessment Sublingual microcirculation will be assessed using the CytoCam-IDF camera (Braedius Medical, Huizen, The Netherlands). The measurement technique involves gently applying the microscope probe with a disposable cap to the sublingual mucosa and recording short video sequences. The device utilizes green LED light to visualize moving blood cells, allowing for subsequent computerized analysis of capillary density and flow quality within the microvessels. Two operators will perform 3 series of measurements at 5-minute intervals with Cytocam - IDF microcirculation camera. Each series will consist of measurements taken from 3 adjacent sites. All measurements will be performed by the same two individuals
  Unit of measurement: mm/mm^2
PVD (Perfused Vessel Density) | From enrollment every 5 minutes (3 measurements per operator) - approx. 20 min.
  Sublingual Microcirculation Assessment Sublingual microcirculation will be assessed using the CytoCam-IDF camera (Braedius Medical, Huizen, The Netherlands). The measurement technique involves gently applying the microscope probe with a disposable cap to the sublingual mucosa and recording short video sequences. The device utilizes green LED light to visualize moving blood cells, allowing for subsequent computerized analysis of capillary density and flow quality within the microvessels. Two operators will perform 3 series of measurements at 5-minute intervals with Cytocam - IDF microcirculation camera. Each series will consist of measurements taken from 3 adjacent sites. All measurements will be performed Unit of measurement: mm/mm^2
PPV (Proportion of Perfused Vessels) | From enrollment every 5 minutes (3 measurements per operator) - approx. 20 min.
  Sublingual Microcirculation Assessment Sublingual microcirculation will be assessed using the CytoCam-IDF camera (Braedius Medical, Huizen, The Netherlands). The measurement technique involves gently applying the microscope probe with a disposable cap to the sublingual mucosa and recording short video sequences. The device utilizes green LED light to visualize moving blood cells, allowing for subsequent computerized analysis of capillary density and flow quality within the microvessels. Two operators will perform 3 series of measurements at 5-minute intervals with Cytocam - IDF microcirculation camera. Each series will consist of measurements taken from 3 adjacent sites. All measurements will be performed by the same two individuals
  Unit of measurement: %
RBCv (Red Blood Cell Velocity) | From enrollment every 5 minutes (3 measurements per operator) - approx. 20 min.
  Sublingual Microcirculation Assessment Sublingual microcirculation will be assessed using the CytoCam-IDF camera (Braedius Medical, Huizen, The Netherlands). The measurement technique involves gently applying the microscope probe with a disposable cap to the sublingual mucosa and recording short video sequences. The device utilizes green LED light to visualize moving blood cells, allowing for subsequent computerized analysis of capillary density and flow quality within the microvessels. Two operators will perform 3 series of measurements at 5-minute intervals with Cytocam - IDF microcirculation camera. Each series will consist of measurements taken from 3 adjacent sites. All measurements will be performed by the same two individuals
  Unit of measurement: mm/s
Heart rate and its variability (HRV) | From enrollment every 5 minutes (3 measurements per operator) - approx. 20 min.
  Heart rate and its variability (HRV) will be recorded using a Holter ECG monitor - electrodes on the chest. Frequency domain method will be used. The number of NN (beat to beat) intervals that match high frequency band (0.15 to 0.4 Hz) or low frequency band (0.04 to 0.15 Hz) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Karol P. Steckiewicz, MD, PhD, Principal Investigator — Medical University of Gdansk; Radosław Owczuk, MD, PhD, DSc, Prof., Principal Investigator — Medical University of Gdansk
Locations (1):
- Medical University of Gdanks, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No